CLINICAL TRIAL: NCT06735690
Title: Pilot/Feasibility Study of CMV-Specific CD19-CAR T Cells Plus CMV-MVA Triplex Following Matched Related Allogeneic Hematopoietic Cell Transplantation for Patients With High-Risk Acute Lymphoblastic Leukemia
Brief Title: Allogeneic CMV-Specific CD19-CAR T Cells Plus CMV-MVA Triplex Vaccine After Matched Related Donor Hematopoietic Cell Transplant for the Treatment of Patients With High-Risk Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24431; NCI-2024-10005 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24431 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Stem Cell Transplantation; Specimen Handling; Biopsy; Leukapheresis; Spinal Puncture; Magnetic Resonance Spectroscopy; Transplantation Conditioning; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (allo CMV-specific CD19-CAR T cells (Experimental): Patients receive HSCT conditioning regimen followed by alloHSCT per standard of care. Starting 28-49 days after alloHSCT, patients receive allo CMV-specific CD19-CAR T cells IV over 10-15 minutes on day 0. Patients undergo ECHO or MUGA, blood and optional CSF sample collection and bone marrow biopsy and aspiration throughout the study. Patient may also undergo chest x-ray and lumbar puncture as needed per PI discretion and PET/CT or CT as clinically indicated throughout the study. Additionally, patients with neurological abnormalities at baseline may undergo MRI of brain throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-CD19-CAR CMV-specific T-lymphocytes; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Leukapheresis; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Other: Transplant Conditioning; Procedure: X-Ray Imaging
- Part 2 (allo CMV-specific CD19-CAR T cells, CMV-MVA vaccine) (Experimental): Patients receive HSCT conditioning regimen followed by alloHSCT per standard of care. Starting 28-49 days after alloHSCT, patients receive allo CMV-specific CD19-CAR T cells IV over 10-15 minutes on day 0. Patients receive CMV-MVA triplex vaccine IM on day 28 in the absence of DLTs and may receive an additional CMV-MVA triplex vaccine IM on day 56 in the absence of DLTs during the second evaluation period. Patients undergo ECHO or MUGA, blood and optional CSF sample collection and bone marrow biopsy and aspiration throughout the study. Patient may also undergo chest x-ray and lumbar puncture as needed per PI discretion and PET/CT or CT as clinically indicated throughout the study. Additionally, patients with neurological abnormalities at baseline may undergo MRI of brain throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-CD19-CAR CMV-specific T-lymphocytes; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Leukapheresis; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Other: Transplant Conditioning; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo alloHSCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Biological: Anti-CD19-CAR CMV-specific T-lymphocytes — Given IV
  Other Names: Anti-CD19-CAR CMV-specific T-cells; CMV-specific CD19 CAR-T Cells; CMV-specific CD19-CAR T Cells
Procedure: Biospecimen Collection — Undergo blood and optional CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given IM
  Other Names: CMV-MVA Triplex Vaccine; Multi-antigen CMV-Modified Vaccinia Ankara Vaccine
  Arms: Part 2 (allo CMV-specific CD19-CAR T cells, CMV-MVA vaccine)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Transplant Conditioning — Given HSCT conditioning regimen
  Other Names: conditioning regimen
Procedure: X-Ray Imaging — Undergo chest x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This early phase I trial tests the safety and side effects of allogeneic CMV-specific CD19-CAR T cells plus CMV-MVA vaccine and how well it works in treating patients with high-risk acute lymphoblastic leukemia after a matched related donor (allogeneic) hematopoietic stem cell transplant (alloHSCT). Chimeric antigen receptor (CAR) T-cell therapy is a type of treatment in which T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood, in this study, the T cells are cytomegalovirus (CMV) specific. Then the gene for a special receptor that binds to a certain protein, CD19, on the patient's cancer cells is added to the CMV-specific T cells in the laboratory. The special receptor is called a CAR. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Vaccines made from three CMV tumor associated antigens, may help the body build an effective immune response to kill cancer cells. Giving allogeneic CMV-specific CD19-CAR T cells plus CMV-MVA vaccine after matched related alloHSCT may be safe, tolerable, and/or effective in treating patients with high-risk acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety and describe the toxicity profile of allogeneic anti-CD19-CAR CMV-specific T-lymphocytes (CMV-specific CD19-CAR T cells) (allo CMV-specific CD19-CAR T cells) alone and when given in combination with multi-peptide CMV-modified vaccinia ankara vaccine (CMV-MVA) triplex vaccine following allogeneic hematopoietic cell transplantation (alloHSCT) to treat participants with high-risk acute lymphoblastic leukemia (ALL).

SECONDARY OBJECTIVES:

I. Determine the feasibility of allo CMV-specific CD19-CAR T cell manufacturing, as assessed by the ability to meet the required cell dose and product release requirements.

II. Estimate the rate of CMV reactivation after CAR T cell infusion with 100 days of HSCT.

III. Estimate the incidence of secondary graft failure. IV. Estimate the incidence and severity of acute graft versus host disease (GVHD) at 100 days and chronic GVHD at 1 year after transplant.

V. Estimate the rate of 100 day non-relapse mortality. VI. Estimate disease-free and overall survival (DFS/OS) rate at 12 months post alloHSCT.

EXPLORATORY OBJECTIVES:

I. Determine short and longer-term allo CMV-specific CD19-CAR T cell expansion and persistence; II. Assess whether the allo CMV-specific CD19-CAR T cells respond to CMV-MVA triplex vaccine III. Assess whether the allo CMV-specific CD19-CAR T cells respond to CMV-MVA triplex vaccine when administered to participants that received CAR T cells only in the safety lead-in portion in the expansion phased of the study (i.e., once safety of the CMV-MVA triplex vaccine is established in the feasibility portion of the study).

OUTLINE:

DONORS: Donors undergo leukapheresis over 2-4 hours.

PART 1: Patients receive HSCT conditioning regimen followed by alloHSCT per standard of care. Starting 28-49 days after alloHSCT, patients receive allo CMV-specific CD19-CAR T cells intravenously (IV) over 10-15 minutes on day 0. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA), blood and optional cerebrospinal fluid (CSF) sample collection and bone marrow biopsy and aspiration throughout the study. Patient may also undergo chest x-ray and lumbar puncture as needed per principal investigator (PI) discretion and positron emission tomography (PET)/computed tomography (CT) or CT as clinically indicated throughout the study. Additionally, patients with neurological abnormalities at baseline may undergo MRI of brain throughout the study.

PART 2: This is a dose-escalation study of followed by a dose-expansion study.

Patients receive HSCT conditioning regimen followed by alloHSCT per standard of care. Starting 28-49 days after alloHSCT, patients receive allo CMV-specific CD19-CAR T cells IV over 10-15 minutes on day 0. Patients receive CMV-MVA triplex vaccine intramuscularly (IM) on day 28 in the absence of DLTs and may receive an additional CMV-MVA triplex vaccine IM on day 56 in the absence of DLTs during the second evaluation period. Patients undergo ECHO or MUGA, blood and optional CSF sample collection and bone marrow biopsy and aspiration throughout the study. Patient may also undergo chest x-ray and lumbar puncture as needed per PI discretion and PET/CT or CT as clinically indicated throughout the study. Additionally, patients with neurological abnormalities at baseline may undergo MRI of brain throughout the study.

After completion of study treatment, patients are followed up monthly for the first year, then at 18, 24, 30 and 36 months after CAR T cell infusion. Patients are then followed up yearly for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study PI approval
* Note: For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated full consent is processed
* Age: ≥ 18 years
* Karnofsky performance status (KPS) ≥ 70
* Participants with high-risk ALL defined as:

  * Any complete remission (CR) with minimal residual disease (MRD)+ (by flow cytometry, polymerase chain reaction [PCR] or clonoSEQ) at the time of HSCT; or
  * Blasts ≥ 5% at the time of transplant; or
  * Complete response (CR)2 or higher irrespective of MRD status; or
  * Requiring > 1 regimen to achieve CR1
* Pathology confirmed CD19+ ALL after the last targeted therapy if the patient has active disease or before the last therapy if the patient is in CR

  * Note: CD19 positivity must be documented in a pathology report; however, it is not a requirement that the CD19 testing be performed by a COH pathologist
* Planned allogeneic HSCT (myeloablative or reduced intensity conditioning) according to institutional eligibility requirements with an available 8/8 (HLA A, B, C, DR) allele-matched related is allowed per discretion of the principal investigator. for allogeneic HSCT will be unmanipulated mobilized peripheral blood stem cell (PBSC) or bone marrow
* Participants who received other prior forms of CAR T therapy are eligible
* No known contraindications to HSCT, leukapheresis, steroids or tocilizum,ab, smallpox vaccine and any other modified vaccinia ankara virus (MVA)-based vaccines
* Total serum bilirubin ≤ 2.0 mg/dL (to be performed no more than 45-days prior to hematopoeitic stem cell [HSC] infusion unless otherwise stated)
* Participants with Gilbert syndrome may be included if their total bilirubin is ≤ 3.0 (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN) (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Alanine aminotransferase < 2.5 x ULN (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Serum creatinine ≤ 2.5 x ULN or estimated creatinine clearance of ≥ 40 mL/min per the Cockcroft-Gault formula, and the participant is not on hemodialysis (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Cardiac function (12 lead-electrocardiogram [ECG]): Corrected QT interval (QTc) must be ≤ 480 msec (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Left ventricular ejection fraction ≥ 45% within 8 weeks before protocol therapy (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Oxygen (O2) saturation > 92% without requiring supplemental oxygen (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Seronegative for HIV quantitative real time polymerase chain reaction (qPCR), hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (RPR) (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed OR
  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
* Negative for COVID-19 within 72 hours of day 0 of protocol therapy (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Negative for human herpes virus-6 (HHV6) by PCR-based assay (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Meets other institutional and federal requirements for infectious disease titer requirements (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)
* Participants must have negative QuantiFERON-TB Gold (QFTG) test (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)

  * Participants with positive QFTG test need clearance from ID before protocol therapy
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test (to be performed no more than 45-days prior to HSC infusion unless otherwise stated)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* DONOR CRITERIA: The identified donor must be the original donor whose stem cells were used for the research participant's alloHSCT
* DONOR CRITERIA: Donor must be CMV seropositive through the following:

  * CMV seropositive AND
  * CMV positive by CMV insight T cell immunity testing through Viracor (Test code 30360)
* DONOR CRITERIA: The donor's hepatitis B surface antigen must be negative and the hepatitis C antibody must be nonreactive. In the case of a positive hepatitis C antibody result, the HCV viral PCR will have to be performed and the results should be negative
* DONOR CRITERIA: The donor must be HIV negative
* DONOR CRITERIA: KPS ≥ 70
* DONOR CRITERIA: Documented body weight
* DONOR CRITERIA: Willingness to sign 'donor consent form' and undergo T cell leukapheresis for the collection of PBMCs for cellular manufacture
* DONOR CRITERIA: COH standard operating procedures (SOP) will be used for allogeneic donor evaluation, selection, and consent.
* DONOR CRITERIA: The donor is approved and has completed the donor evaluation per institutional guidelines. Additionally, donor will also be screened for the following infectious diseases:

  * Epstein-Barr virus (EBV) by PCR,
  * Human herpes virus 6, 7, and 8 (HHV6, HHV7, HHV8)
  * Parvovirus B19 Note: ID test results for EBV by PCR, HHV6, HHV7, HHV8 and parvovirus B19 are necessary to proceed with the apheresis procedure but do have to be resulted and negative before participant CAR T infusion.

Donor screening will be in compliance with all requirements of Food and Drug Administration (FDA) regulation 21 CFR Part 1271 including donor screening for COVID-19 exposure or infection.

Exclusion Criteria:

* Concurrent use of systemic steroids. Recent or current use of inhaled or topical steroids in standard doses is not exclusionary. Physiologic replacement of steroids (prednisone ≤ 0.5 mg /day, or equivalent doses of other corticosteroids) is allowed
* Participants with active autoimmune disease requiring systemic immune suppressive therapy are not allowed
* Any contraindications to standard conditioning transplant regimens per standard of care practices at COH
* Subjects with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of screening
* History or prior diagnosis of other immunologic or inflammatory disease affecting the central nervous system (CNS), including uncontrolled seizure disorder, any measurable masses of CNS, or any other active CNS disease. Note: Research participants with a history of CNS disease that has been effectively treated to complete remission (< 5 white blood cells [WBC]/mm^3 and no blasts in CSF) will be eligible
* Participants should not have any uncontrolled illness including symptomatic congestive heart failure, unstable angina pectoris, poorly controlled pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* History of stroke or intracranial hemorrhage within 3 months prior to screening
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* Participants with uncontrolled seizures
* Active viral hepatitis
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; non-muscle invasive bladder cancer; malignancy treated with curative intent with no known active disease present for ≥ 2 years
* Clinically significant uncontrolled illness
* Active infection not responding to antibiotics
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2029-03-07 (Estimated); Study Completion 2029-03-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  Will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. AEs will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Dose-limiting toxicities (DLT) | Up to 28 days after T cell infusion
  Will be graded according to NCI CTCAE v 5.0, and the revised American Society for Transplantation and Cellular Therapy Cytokine Release Syndrome Cytokine Release Syndrome grading system.

SECONDARY OUTCOMES:
Achieving required cell dose and product release requirements | Up to first segment of the trial (6 weeks)
Disease status | At days 0 and 72 and months 5 and 11
  Will be evaluated based on grading of tumor responses according to the National Comprehensive Cancer Network Clinical Practice Guidelines in Oncology for acute lymphoblastic leukemia. Will be assessed using linear mixed effects modeling. The overall fit of the model will be evaluated graphically by taking a scatter plot of data for the chimeric antigen receptor (CAR) T cells and applying an overlay of the line generated by the model. To assess changes over time, functional regression modeling will be used. Similar modeling techniques will be used to assess the impact of combination treatment (CAR T cells and vaccine) on clinical events (e.g., disease response). Swimmer plots will be generated to show response status after infusion of CAR T cells, vaccination, DLTs, and other clinical outcomes such as disease progression or death of each participant.
Secondary graft failure | Up to 15 years
  Will be defined as loss of donor cells after initial engraftment. Graft failure is defined as > 95% recipient CD3+ or CD34+ cells at any single time after engraftment in the absence of leukemia relapse.
Cytomegalovirus reactivation requiring antiviral treatment | Up to 100 days after transplant
  Will be assessed using polymerase chain reaction.
Acute graft versus host disease (GVHD) | From date of stem cell infusion to documented/biopsy proven acute GVHD onset date, assessed up 100 days
  Will assessed and graded according to the Mount Sinai Acute GVHD International Consortium grading. Cumulative incidence will be estimated.
Chronic GVHD | From approximately 80-100 days post-transplant to the documented/biopsy proven chronic GVHD onset date, assessed at 1 year
  Will be scored according to the National Institute of Health Consensus staging. Cumulative incidence will be estimated.
Non-relapse mortality (NRM) | From start of protocol therapy until non-disease related death, or last follow up, whichever comes first, assessed at 100 days
  NRM is calculated using the Fine and Gray method as a competing risk with disease relapse.
Disease-free survival | From the start of protocol therapy to the date of death, disease relapse, or last follow-up whichever occurs first, assessed at 1 year
  Will be estimated using the product-limit method of Kaplan-Meier.
Overall survival | From start of protocol therapy to death, or last follow-up, whichever occurs first, assessed at 1 year
  Will be estimated using the product-limit method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Aldoss, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States